CLINICAL TRIAL: NCT00530491
Title: Prospective Randomized Controlled Trial to Reduce Morbidity and Mortality After Lung Surgery in Patients With FEV1 < 70% of Expected Value or < 1.5L
Brief Title: Prospective Trial to Reduce Morbidity and Mortality After Lung Surgery in Patients With Reduced Pulmonary Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Bernd Muehling, M.D., Dep. of Thoracic and Vascular Surgery, University of Ulm , Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BM 140/07
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2008-02-14 (Estimated); Status verified 2007-09

CONDITIONS: Respiration Disorders
Keywords: lung resection; reduced pulmonary function
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): conventional perioperative management for lung surgery
  Interventions: Procedure: Fast track lung surgery
- 2 (Experimental): fast track management for lung surgery
  Interventions: Procedure: Fast track lung surgery

INTERVENTIONS:
Procedure: Fast track lung surgery — fast track lung surgery: carbohydrate drink preoperatively, PCEA, early removal of chest tube conventional: no carbohydrate drink preoperatively, ICB+PCA, removal of chest tube depending upon chest x-ray

SUMMARY:
A fast track recovery program (thoracic epidural anesthesia, carbohydrate drink preoperative, early removal of chest tubes) is evaluated compared to conventional perioperative treatment (patient controlled analgesia, no carbohydrate drink preoperative) in patients with FEV1 < 70% of expected value or < 1.5L who undergo resections of the lung.

ELIGIBILITY:
Inclusion Criteria:

* resection of the lung
* FEV1 <70% of expected value or below 1.5L
* 18-80y
* given written informed consent

Exclusion Criteria:

* contraindication for epidural anesthesia
* prio ipsilateral thoracotomy
* chemotherapy <6 weeks prior to study enter
* existing pneumonia (fever, elevated WCC, elevated CRP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
pulmonary complications (air leak, atelectasis, pneumonia); lung function on pod 7; overall mortality | 1 year

SECONDARY OUTCOMES:
duration of ICU treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bernd M Muehling, M.D., Study Chair
Locations (1):
- University of Ulm, Ulm, Germany